CLINICAL TRIAL: NCT00188981
Title: Dutch Prediction of Psychosis Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Other Study IDs: CCMOP02.0441C; METC02/178
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Psychotic Disorders
Keywords: psychosis; high risk; prodrome; Multiple Complex Developmental Disorder
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The Dutch Prediction of Psychosis Study (DUPS) is a prospective study of predictors of the transition to psychosis in help-seeking adolescents at high risk for developing a first psychotic episode. The aim of the project is supplemented by a systematic account of the pathways to care, the disabilities and needs and the therapeutic interventions that are currently used in this population.

Multi-level assessment includes behavioral and cognitive variables as well as structural brain imaging and neurophysiological data. Subjects will be followed up at regular intervals during (at least) two years to monitor the development of their (psychotic) symptoms. This will allow us to analyze the predictive validity of the variables.

DETAILED DESCRIPTION:
The Dutch Prediction of Psychosis Study (DUPS) is a collaboration of the Academic Medical Center in Amsterdam (AMC) and the University Medical Center in Utrecht (UMC). The main objectives are:

1. Pathways to care: the description of the ways subjects at risk for psychosis get access to the health care system and the detection of obstacles to adequate treatment
2. Prediction: the systematic multi-level assessment of predictors of the transition to a first psychotic episode in subjects at risk for psychosis
3. Disability: the description of disabilities, deficits and needs in prodromal individuals
4. Intervention: the description of the therapeutic and preventive interventions applied to prodromal individuals

While the same fundamental principles (e.g. inclusion criteria) are applied in both centers, additional instruments or paradigms are added in the separate centers according to specific interests, expertise and setting.

Our specific interest is in the social cognition and social functioning of prepsychotic individuals. Therefore, in addition to the subjects that are at high risk for psychosis according to the DUPS inclusion/exclusion criteria we are including another group of subjects that is at elevated risk for psychosis, namely subjects who have a Multiple Complex Developmental Disorder (MCDD) which is a subtype of the pervasive developmental disorders.

The study is a prospective longitudinal field-study with repeated measures to monitor subjects at high risk for psychosis.

The study sample in the UMC consists of adolescents who are already referred to adolescent psychiatric outpatient's clinics because of mental problems. After informed consent they are screened for the following inclusion and exclusion criteria:

1. Age between 12 and 18 years
2. No previous psychotic episode for more than one week
3. Verbal IQ above 75
4. Symptoms are not due to an organic mental disorder or substance abuse
5. Belong to one or more of the following groups:

   1. Basic symptoms: presence of self-perceived cognitive thought disturbances
   2. Familial risk plus reduced functioning: having a first- or second degree relative with a history of any psychotic disorder in combination with a deterioration of mental state and/or social functioning in the last year
   3. Attenuated psychotic symptoms: presence of psychotic symptoms at sub-clinical level
   4. Brief, limited or intermittent psychotic symptoms: having a history of psychotic symptoms with a duration of less than one week and spontaneous remission
   5. Multiple Complex Developmental Disorder

Assessment includes:

1. basic clinical assessment
2. neuropsychological measures (attention, memory, executive functioning)
3. social cognitive measures (facial emotion recognition, mentalizing, social attribution)
4. measures of social cognition and behavior
5. EEG and Event Related Potentials (including smooth pursuit eye movement, auditory mismatch negativity)
6. structural MRI

Some data will be collected retrospectively upon inclusion into the study, for example symptom history and pathways to care. Outcome is assessed after 9, 18 and 24 months.

ELIGIBILITY:
Inclusion criteria:

Help-seeking adolescents who belong to one or more of the following groups:

* Basic symptoms: presence of self-perceived cognitive thought disturbances
* Familial risk plus reduced functioning: having a first- or second degree relative with a history of any psychotic disorder in combination with a deterioration of mental state and/or social functioning in the last year
* Attenuated psychotic symptoms: presence of psychotic symptoms at sub-clinical level
* Brief, limited or intermittent psychotic symptoms: having a history of psychotic symptoms with a duration of less than one week and spontaneous remission
* Multiple Complex Developmental disorder

Exclusion criteria:

* A previous psychotic episode for more than one week
* Verbal IQ < 75
* Symptoms are due to an organic mental disorder or substance abuse

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2003-06; Study Completion 2008-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Schothorst, PhD, Principal Investigator — University Medical Center Utrecht, department of Child and Adolescent Psychiatry; Herman van Engeland, Professor, Principal Investigator — University Medical Center Utrecht, department of Child and Adolescent Psychiatry
Locations (1):
- University Medical Center Utrecht, department of Child and Adolescent Psychiatry, Utrecht, Utrecht, Netherlands